CLINICAL TRIAL: NCT02448901
Title: Influence of Edoxaban on Coagulability and Thrombin Generation: An in Vitro Study Focusing on Thrombelastography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, Paul A. Gurbel, Director, Sinai Center for Thrombosis Research, LifeBridge Health
Other Study IDs: 2213
Record Dates: First submitted 2015-04-23; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Edoxaban — In vitro study. Various concentrations of Edoxoban added to blood sample and tested
  Other Names: DU-176b, trade names Savaysa, Lixiana

SUMMARY:
The influence of different doses of edoxaban on physical characteristics of the clot and thrombin generation kinetics in blood samples will be studied by in vitro spiking of blood samples collected from patients treated for heart failure (with and without hypercoagulability) and from healthy volunteers (with and without hypercoagulability). This in vitro experiment will help us to:

(i) detect qualitative anticlotting properties of edoxaban. (ii) quantify the anticlotting properties of edoxaban.

DETAILED DESCRIPTION:
Experimental protocol

1. On the day of experiment blood samples will be collected in 3.2% citrate tubes.
2. One citrated blood tube will be centrifuged to collect plasma for biomarker measurements (C-reactive protein (CRP), fibrinogen, von Willebrand factor (vWF), interleukin (IL)-6, p-selectin, plasminogen activator inhibitor (PAI)-1, matrix metalloproteinase (MMP)-9).
3. Blood samples will be incubated with different concentrations of edoxaban (no edoxaban, subtherapeutic range - 30 nM, therapeutic range -300 nM, and supratherapeutic range- 900 nM) (3).

A) Cora® Hemostasis Analyzer System (Cora®) will be used to assess qualitative and quantitative assessment of the hemostatic properties of a blood sample in the presence or absence of edoxaban. The CORA is an integrated computer module with Ethernet connection capability and provides continuous resonance-frequency viscoelasticity measurements using a disposable four-channel microfluidic cartridge to determine simultaneous maximal platelet-fibrin clot strength, fibrin clot strength, and response to antiplatelet agents or anticoagulants. The cartridge has four channels - citrated Kaolin (CK) channel that measures platelet-fibrin clot strength, anti-Xa channel, DTI channel and FFC channel that measures contribution of functional fibrinogen.

In addition, using the V-curve software, the following parameters of thrombin generation kinetics will be evaluated from the CK channel- R - Period of time of latency from the time that the blood was placed in the TEG® analyzer until the initial fibrin formation. This represents the enzymatic portion of coagulation.

K - K time is a measure of the speed to reach a certain level of clot strength. This represents clot kinetics.

alpha - measures the rapidity of fibrin build-up and cross-linking (clot strengthening). This represents fibrinogen level.

MA - Maximum Amplitude is a direct function of the maximum dynamic properties of fibrin and platelet bonding via GPIIb/IIIa and represents the ultimate strength of the fibrin clot. This represents platelet function/aggregation.

TMRTG - Time to maximum rate of thrombus generation. MRTG - Maximum rate of thrombus generation. TG - Total thrombus generated. TMRL - Time to maximum rate of lysis MRL - Maximum rate of lysis L - Total lysis D - Delta is the difference between R time and the time of initial split point (SP, mins) of the TEG tracing (R - SP), representing the time interval of greatest clot growth secondary to peak thrombin generation.

B) Calibrated Automated Thrombogram® (CAT) System: Lag time, peak thrombin production, mean velocity rate index and endogenous thrombin potential (ETP) will be assessed by calibrated automated thrombogram in platelet poor plasma (Thrombinoscope by Stago).

ELIGIBILITY:
Inclusion Criteria:

Patients with heart failure (class I-IV) are eligible for enrollment:

1. Patient must have documented symptomatic chronic HF for at least 3 months prior to screening. Exacerbation of chronic HF is defined as symptoms of worsening dyspnea or fatigue, objective signs of congestion such as peripheral edema or ascites, and/or adjustment of pre-hospitalization HF medications.
2. Subject must have a documented LVEF of less than or equal to 40% within 3 months of the study. If more than one LVEF is available, the most recent one should be used, but it must be less than or equal to 40%. The ejection fraction will be determined by one of the following methods: echocardiogram, nuclear multigated acquisition (MUGA) scan, cardiac MRI, cardiac CT scan, or left ventriculography.
3. Patient must be receiving appropriate HF treatment at the appropriate dosing per guidelines:

   * Diuretic (required for study entry) Renin-angiotensin system (RAS) inhibitors such as an ACE inhibitor, or ARB if intolerant of ACE inhibitor, or vasodilator therapy such as hydralazine or nitrates if intolerant to ACE inhibitor and ARB
   * Beta blocker therapy
   * Aldosterone antagonist therapy.
4. Patient must have completed all prophylactic anticoagulation (such as enoxaparin, warfarin, heparin, etc) for at least one week before study.
5. Each patient (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and is willing to participate in the study.

Exclusion Criteria:

For Healthy Subjects:

subjects currently on antiplatelet therapy or any other agents that are known to influence platelet function and coagulation.

For Subjects with Heart Failure:

1. Hemodynamic instability, active bleeding and bleeding diatheses, oral anticoagulation therapy, leukocyte count < 3,000/mm3, platelet count < 100,000/mm3, aspartate aminotransferase or alanine aminotransferase levels ≥ 3 times upper normal, and creatinine >2mg/dL.
2. Patient has a severe concomitant disease such as: Atrial fibrillation (AFib) or another condition that requires chronic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers (n=20) Heart Failure Patients (n=20)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of clot physiology of a blood sample in the presence and absence of edoxaban by point of care thrombelastography (TEG-6s) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: paul gurbel, MD, Principal Investigator — Sinai Center for Thrombosis Research
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States